CLINICAL TRIAL: NCT00468819
Title: Open-label Multi-center Study of Magnetic Resonance Imaging (MRI) With 0.1 mmol/kg Body Weight (BW) Gadavist (1.0 M) to Assess Pharmacokinetics, Safety and Tolerability in Children.
Brief Title: A Study of Magnetic Resonance Imaging (MRI) With Gadavist in Children
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 91552; 2006-004153-22 (EudraCT Number); 310788 (Other: Company internal)
Record Dates: First submitted 2007-05-02; First posted 2007-05-03 (Estimated); Results first posted 2011-09-05 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-06

CONDITIONS: Magnetic Resonance Imaging
Keywords: Contrast-enhanced MRI; MR angiography (MRA) Children 2-17 years
MeSH Terms: interventions — gadobutrol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Gadobutrol (Gadavist, BAY86-4875) - age 2 to 6 years (Experimental): Participants received Gadobutrol 0.1 mmol/kg body weight (BW) = 0.1 mL/kg BW as single intravenous bolus injection
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875)
- Gadobutrol (Gadavist, BAY86-4875) - age 7 to 11 years (Experimental): Participants received Gadobutrol 0.1 mmol/kg body weight (BW) = 0.1 mL/kg BW as single intravenous bolus injection
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875)
- Gadobutrol (Gadavist, BAY86-4875) - age 12 to 17 years (Experimental): Participants received Gadobutrol 0.1 mmol/kg body weight (BW) = 0.1 mL/kg BW as single intravenous bolus injection
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875)
- Gadobutrol (Gadavist, BAY86-4875) - age 2 to 17 years (Experimental): Participants received Gadobutrol 0.1 mmol/kg body weight (BW) = 0.1 mL/kg BW as single intravenous bolus injection
  Interventions: Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875)

INTERVENTIONS:
Drug: Gadobutrol (Gadavist, Gadovist, BAY86-4875) — In an open-label design, all patients will receive a total dose of 0.1 mmol/kg BW Gadovist 1.01 Days Injection

SUMMARY:
In this clinical study a contrast agent for magnetic resonance imaging (MRI), which has already been approved for application in adults, will be investigated in children and adolescents. MRI is a modern and safe examination method without delivering radiation burden using magnetic fields to produce cross-sectional images of the human body. A special computer program then puts these images together and creates a two or three-dimensional image of the inner organs thus facilitating the detection and evaluation of pathological changes. In contrast-enhanced MRI a contrast agent is injected into a peripheral vein before the examination which results in a stronger contrast in the examined area. Therefore, pathological changes can be more easily detected and evaluated compared to non-enhanced MRI. The company Bayer HealthCare Pharmaceuticals has developed a contrast agent for MRI called Gadavist 1.0 which was first approved in 1998 in Switzerland for MRI of brain and spine. Since 2003 Gadavist can also be used in magnetic resonance angiography (MRA) in adults, i.e. in the MRI examination of the blood vessels and since 2006 in MRI of liver and kidney disease. Gadavist was examined in more than 2,900 adults within the framework of clinical studies during development and has been used after its marketing authorization in meanwhile more than 600,000 patients. Yet, clinical studies investigating Gadavist have been only conducted with adults so far. Diseases requiring MRI examinations, however, often occur in children, too. Therefore, many contrast agents are already used on a regular basis in MRI examinations of children, some of these contrast agents being authorized already. Within the framework of this study the pharmacokinetic characteristics of Gadavist in children or adolescents will be investigated, i.e. how the contrast agent is distributed and behaves in the body. In addition, safety and tolerability will be evaluated in order to demonstrate that Gadavist 1.0 is a safe and well tolerated contrast agent also for children and adolescents. Furthermore, the study aims to obtain the dosage recommendation of 0.1 ml per kilogram body weight also for this population group.

DETAILED DESCRIPTION:
Please note that the present study is allocated two study phases, i.e. phase I and phase III.

ELIGIBILITY:
Inclusion Criteria:

* Patients (male/ female) of specific age groups (2-6 years, 7-11 years, 12-17 years) who are scheduled to undergo Gadolinium (Gd)-enhanced MRI of brain, spine, liver and/or kidneys or Gd-enhanced MRA (single field of view).

Exclusion Criteria:

* Clinically unstable patients (e.g. intensive care unit)
* Renal insufficiency
* Patients undergoing a relevant change in chemotherapy </= 48 hours prior to and up to 24 hours after the administration of Gadovist.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 140 (Actual)
Dates: Start 2007-05; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (13):
- Vienna, Vienna, Austria
- Canada (2):
  - Edmonton, Alberta
  - Toronto, Ontario
- Germany (7):
  - Erlangen, Bavaria
  - Bonn, North Rhine-Westphalia
  - Dresden, Saxony
  - Leipzig, Saxony
  - Halle, Saxony-Anhalt
  - Kiel, Schleswig-Holstein
  - Jena, Thuringia
- Sweden (3):
  - Gothenburg
  - Stockholm
  - Uppsala

REFERENCES:
- [Result] Hahn G, Sorge I, Gruhn B, Glutig K, Hirsch W, Bhargava R, Furtner J, Born M, Schroder C, Ahlstrom H, Kaiser S, Moritz JD, Kunze CW, Shroff M, Stokland E, Trnkova ZJ, Schultze-Mosgau M, Reif S, Bacher-Stier C, Mentzel HJ. Pharmacokinetics and safety of gadobutrol-enhanced magnetic resonance imaging in pediatric patients. Invest Radiol. 2009 Dec;44(12):776-83. doi: 10.1097/RLI.0b013e3181bfe2d2. PMID 19858730
- [Result] Reif S, Schultze-Mosgau M, Sutter G. From adults to children: simulation-based choice of an appropriate sparse-sampling schedule. Paediatr Drugs. 2012 Jun 1;14(3):189-200. doi: 10.2165/11595430-000000000-00000. PMID 22409261
- See also: Click here to find information about studies related to Bayer Healthcare products conducted in Europe — http://www.clinicaltrialsregister.eu/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years
Started | 48 (Enrolled participants) | 44 (Enrolled participants) | 48 (Enrolled participants)
Treatment Received/ Safety Follow-up | 46 (FAS (Full Analysis Set)) | 44 (FAS) | 48 (FAS)
Completed | 42 | 44 | 46
Not Completed | 6 | 0 | 2
Not completed — Withdrawal by Subject | 4 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Drop-outs (Treatment never received) | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Total
Number analyzed (Participants) | 46 | 44 | 48 | 138
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.7 (1.46) | 9.0 (1.38) | 14.7 (1.80) | 9.2 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 13 | 23 | 53
  Male | 29 | 31 | 25 | 85
Body Weight [Mean (Standard Deviation); unit: kg] | 17.49 (5.434) | 33.75 (8.956) | 57.19 (14.245) | 36.48 (19.447)

OUTCOME MEASURES:

1. Primary Outcome: Plasma Clearance Estimates of Gadobutrol by Age Group
Description: Total body clearance of Gadobutrol in plasma in L/h after intravenous injection.
Time Frame: From injection of Gadobutrol up to 8 hours after injection.
Population: Final pharmacokinetics (PK) analysis set
Measure: Median (Inter-Quartile Range); unit: L/h
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 45 | 39 | 46 | 130
L/h | 2.07 [1.45 to 3.83] | 3.28 [1.81 to 5.93] | 4.90 [2.52 to 7.37] | 3.24 [1.53 to 6.62]

2. Primary Outcome: Body Weight-corrected Plasma Clearance Estimates of Gadobutrol by Age Group
Description: Total body clearance of Gadobutrol in plasma corrected for body weight (L/h/kg) after intravenous injection.
Time Frame: From injection up to 8 hours after Gadobutrol injection
Population: Final PK analysis set
Measure: Median (Inter-Quartile Range); unit: L/h/kg
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 45 | 39 | 46 | 130
L/h/kg | 0.13 [0.09 to 0.17] | 0.10 [0.05 to 0.17] | 0.09 [0.05 to 0.10] | 0.10 [0.05 to 0.17]

3. Primary Outcome: Volume Distribution at Steady State (Vss) Estimates of Gadobutrol by Age Group
Description: Apparent volume of distribution at steady state expressed in L after intravenous injection.
Time Frame: From injection up to 8 hours after Gadobutrol injection
Population: Final PK analysis set
Measure: Median (Inter-Quartile Range); unit: L
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 45 | 39 | 46 | 130
L | 3.83 [3.24 to 6.33] | 5.98 [4.06 to 11.69] | 10.02 [5.16 to 14.12] | 5.96 [3.27 to 13.21]

4. Primary Outcome: Body Weight-corrected Volume Distribution at Steady State (Vss) Estimates of Gadobutrol by Age Group
Description: Apparent volume of distribution at steady state corrected for body weight (L/h/kg) after intravenous injection.
Time Frame: From injection to 8 hours after Gadobutrol injection
Population: Final PK analysis set
Measure: Median (Inter-Quartile Range); unit: L/kg
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 45 | 39 | 46 | 130
L/kg | 0.24 [0.20 to 0.28] | 0.19 [0.14 to 0.23] | 0.18 [0.09 to 0.23] | 0.20 [0.12 to 0.28]

5. Primary Outcome: Area Under the Drug Concentration-time Curve of Gadobutrol by Age Group
Description: Area under the concentration versus time curve from zero to infinity after intravenous injection expressed in µmol*h/L.
Time Frame: From injection to 8 hours after Gadobutrol injection
Population: Final PK analysis set
Measure: Median (Inter-Quartile Range); unit: µmol*h/L
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 45 | 39 | 46 | 130
µmol*h/L | 815 [494 to 1167] | 969 [590 to 2163] | 1167 [925 to 1808] | 999 [590 to 1808]

6. Primary Outcome: Terminal Elimination Half Life Estimates of Gadobutrol by Age Group
Description: Terminal elimination half-life of Gadobutrol from plasma expressed in h and derived from the terminal slope of the concentration versus time curve.
Time Frame: From injection to 8 hours after Gadobutrol injection
Population: Final PK analysis set
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 45 | 39 | 46 | 130
hours | 1.75 [1.34 to 2.30] | 1.61 [1.17 to 2.62] | 1.65 [1.42 to 2.23] | 1.69 [1.34 to 2.32]

7. Primary Outcome: Mean Residence Time (MRT) Estimates of Gadobutrol by Age Group
Description: Mean residence time of Gadobutrol in plasma expressed in h.
Time Frame: From injection to 8 hours after Gadobutrol injection
Population: Final PK analysis set
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 45 | 39 | 46 | 130
hours | 1.88 [1.24 to 2.77] | 1.83 [1.03 to 3.37] | 2.03 [1.57 to 2.99] | 1.94 [1.24 to 2.99]

8. Secondary Outcome: Urinary Excretion of Gadolinium as Percent of Administered Dose
Description: Amount of gadolinium* excreted into urine during the collection interval 0 - 6 h post dose expressed as % of administered dose. *A metallic rare-earth element, used as a contrast medium for magnetic resonance imaging.
Time Frame: up to 6 hours after Gadobutrol injection
Population: Valid for urinary analysis
Measure: Mean (Full Range); unit: percentage of administered dose
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 22 | 34 | 41 | 97
percentage of administered dose | 93.78 [9.19 to 187.73] | 92.14 [18.96 to 117.18] | 95.96 [3.48 to 139.03] | 94.13 [3.48 to 187.73]

9. Secondary Outcome: Number of Participants With Basic Technical Adequacy of Magnetic Resonance (MR) Images for Diagnosis by Age Group
Description: In the participants the technical adequacy (evaluability) of MR images was assessed on the following 4-point scale (1=not adequate [compromised quality], 2=partially adequate [evaluation possible], 3=adequate despite artifacts, 4=adequate with excellent quality).
Time Frame: Up to 1 hour after Gadobutrol injection
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 46 | 44 | 48 | 138
Participants
  not adequate (compromised quality) | 0 | 0 | 1 | 1
  partially adequate (evaluation possible) | 0 | 0 | 0 | 0
  adequate despite artifacts | 12 | 13 | 14 | 39
  adequate with excellent quality | 34 | 31 | 33 | 98

10. Secondary Outcome: Number of Participants With Overall Contrast Quality of Post Contrast Images by Age Group
Description: In the participants qualitative overall contrast quality of post contrast images was assessed on the following 6-point scale (none, poor, moderate, good, excellent, not assessable).
Time Frame: up to 1 hour after Gadobutrol injection
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 46 | 44 | 48 | 138
Participants
  none | 0 | 0 | 0 | 0
  poor | 0 | 0 | 0 | 0
  moderate | 0 | 0 | 3 | 3
  good | 9 | 17 | 13 | 39
  excellent | 37 | 27 | 32 | 96
  not assessable | 0 | 0 | 0 | 0

11. Secondary Outcome: Pre-Contrast Lesions by Location and by Age Group
Description: Number of lesions on pre-contrast images by organ location and age group.
Time Frame: up to 1 hour after Gadobutrol injection
Population: FAS
Measure: Number; unit: Lesions
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 46 | 44 | 48 | 138
Lesions
  Kidney | 5 | 0 | 8 | 13
  Liver | 0 | 0 | 0 | 0
  Brain | 34 | 32 | 30 | 96
  Vessel | 0 | 0 | 0 | 0
  Spine | 7 | 2 | 1 | 10

12. Secondary Outcome: Post-Contrast Lesions by Location and by Age Group
Description: Number of lesions on post-contrast images by organ location and age group.
Time Frame: up to 1 hour after Gadobutrol injection
Population: FAS
Measure: Number; unit: Lesions
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 46 | 44 | 48 | 138
Lesions
  Kidney | 6 | 0 | 5 | 11
  Liver | 0 | 0 | 0 | 0
  Brain | 33 | 32 | 34 | 99
  Vessel | 0 | 0 | 2 | 2
  Spine | 7 | 2 | 1 | 10

13. Secondary Outcome: Pre-Contrast Delineation of Lesion/Vessel Border by Age Group
Description: In the participants pre-contrast delineation of each lesion/vessel border was assessed on the following 5-point scale (no, moderate, good, excellent, not assessable).
Time Frame: up to 1 hour after Gadobutrol injection
Population: FAS
Measure: Number; unit: Lesions
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 46 | 44 | 48 | 138
Lesions
  no | 3 | 0 | 1 | 4
  moderate | 5 | 0 | 5 | 10
  good | 20 | 20 | 15 | 55
  excellent | 18 | 14 | 18 | 50
  not assessable | 0 | 0 | 0 | 0

14. Secondary Outcome: Post-Contrast Delineation of Lesion/Vessel Border by Age Group
Description: In the participants post-contrast delineation of each lesion/vessel border was assessed on the following 5-point scale (no, moderate, good, excellent, not assessable).
Time Frame: up to 1 hour after Gadobutrol injection
Population: FAS
Measure: Number; unit: Lesions
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 46 | 44 | 48 | 138
Lesions
  no | 0 | 0 | 5 | 5
  moderate | 0 | 4 | 7 | 11
  good | 14 | 10 | 10 | 34
  excellent | 30 | 20 | 19 | 69
  not assessable | 2 | 0 | 1 | 3

15. Secondary Outcome: Pre-Contrast Lesion Characterization by Age Group
Description: In the participants the internal morphology and structure of each pre-contrast lesion was assessed on the following 4-point scale (1=poor, 2=moderate, 3=good, 4=not applicable).
Time Frame: up to 1 hour after Gadobutrol injection
Population: FAS
Measure: Number; unit: Lesions
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 46 | 44 | 48 | 138
Lesions
  poor | 3 | 1 | 2 | 6
  moderate | 6 | 6 | 6 | 18
  good | 36 | 27 | 30 | 93
  not applicable | 1 | 0 | 1 | 2

16. Secondary Outcome: Post-Contrast Lesion Characterization by Age Group
Description: In the participants the internal morphology and structure of each post-contrast lesion was assessed on the following 4-point scale (1=poor, 2=moderate, 3=good, 4=not applicable).
Time Frame: up to 1 hour after Gadobutrol injection
Population: FAS
Measure: Number; unit: Lesions
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 46 | 44 | 48 | 138
Lesions
  poor | 1 | 0 | 6 | 7
  moderate | 2 | 3 | 6 | 11
  good | 42 | 31 | 25 | 98
  not applicable | 1 | 0 | 5 | 6

17. Secondary Outcome: Degree of Contrast Enhancement in Lesion/Vessel by Age Group (Given Are Total Numbers of Lesions)
Description: In the participants the degree of contrast enhancement in each lesion/vessel was assessed on the following 5-point scale (1=no, 2=moderate, 3=good, 4=excellent, 5=not applicable).
Time Frame: up to 1 hour after Gadobutrol injection
Population: FAS
Measure: Number; unit: Lesions
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 46 | 44 | 48 | 138
Lesions
  no | 19 | 19 | 18 | 56
  moderate | 1 | 1 | 4 | 6
  good | 3 | 4 | 2 | 9
  excellent | 20 | 10 | 16 | 46
  not applicable | 3 | 0 | 2 | 5

18. Secondary Outcome: Number of Participants With Change in Diagnostic Confidence by Age Group
Description: In the participants the change in diagnostic confidence (additional diagnostic gain by the post-contrast scan) was assessed on the following 3-point scale (1=unchanged, 2=improved, 3=worsened).
Time Frame: up to 1 hour after Gadobutrol injection
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Number analyzed (Participants) | 46 | 44 | 48 | 138
Participants
  missing | 0 | 0 | 1 | 1
  unchanged | 3 | 3 | 5 | 11
  improved | 43 | 41 | 42 | 126
  worsened | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years
Serious Adverse Events (participants affected / at risk) | 1/46 | 1/44 | 0/48 | 2/138
Other Adverse Events (participants affected / at risk) | 17/46 | 16/44 | 16/48 | 49/138
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years (N=46) | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years (N=44) | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years (N=48) | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years (N=138)
Meningitis (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Crystal urine (Investigations) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 6 Years (N=46) | Gadobutrol (Gadavist, BAY86-4875) - Age 7 to 11 Years (N=44) | Gadobutrol (Gadavist, BAY86-4875) - Age 12 to 17 Years (N=48) | Gadobutrol (Gadavist, BAY86-4875) - Age 2 to 17 Years (N=138)
Eosinophilia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 1 | 1 | 3
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Constipation (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Enteritis (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 1 | 3 | 5
Stomach discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Vomiting (Gastrointestinal disorders) | 2 | 2 | 1 | 5
Chest pain (General disorders) | 0 | 1 | 0 | 1
Feeling hot (General disorders) | 0 | 0 | 2 | 2
Pyrexia (General disorders) | 2 | 2 | 1 | 5
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 1
Gastroenteritis (Infections and infestations) | 2 | 1 | 0 | 3
Gastrointestinal infection (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1 | 1 | 2
Otitis media (Infections and infestations) | 1 | 0 | 0 | 1
Rhinitis (Infections and infestations) | 0 | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0 | 2
Central line infection (Infections and infestations) | 1 | 0 | 0 | 1
Oral herpes (Infections and infestations) | 1 | 0 | 0 | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 2 | 2
Headache (Nervous system disorders) | 0 | 2 | 2 | 4
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1
Dysuria (Renal and urinary disorders) | 0 | 0 | 1 | 1
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1 | 1
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1

LIMITATIONS AND CAVEATS:
Originally, urine was collected up to 6 hours post injection in patients > 9 years. This was amended to patients of all age groups. As a result, urine was collected in 102 of 138 patients with gadobutrol injection (lowest rate in patients 2-6 years).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less